CLINICAL TRIAL: NCT01359787
Title: Double-blind, Randomized, Vehicle-controlled, Multicenter, Multinational, Parallel-group Study of the Efficacy and Safety of Mapracorat Ointment in Three Concentrations Over Max. 4 Weeks in Subjects With Atopic Dermatitis (AD)
Brief Title: Efficacy and Safety of Different Concentrations of Mapracorat Ointment Over 4 Weeks in Atopic Dermatitis (AD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15616; 1403440 (Other: Company internal); 2010-024279-14 (EudraCT Number)
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Atopic Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — R-1,1,1-trifluoro-4-(5-fluoro-2,3-dihydrobenzofuran-7-yl)-4-methyl-2-(((2-methyl-5-quinolyl)amino)methyl)pentan-2-ol; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mapracorat 0.01% Ointment (Active Comparator): Lowest concentration
  Interventions: Drug: Mapracorat
- Mapracorat 0.03% Ointment (Active Comparator): Middle concentration
  Interventions: Drug: Mapracorat
- Mapracorat 0.1% Ointment (Active Comparator): Highest concentration
  Interventions: Drug: Mapracorat
- Vehicle without active (Placebo Comparator)
  Interventions: Drug: Vehicle without active

INTERVENTIONS:
Drug: Mapracorat — Daily topical application
  Arms: Mapracorat 0.01% Ointment; Mapracorat 0.03% Ointment; Mapracorat 0.1% Ointment
Drug: Vehicle without active — Daily topical application
  Arms: Vehicle without active

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of three concentrations of a development drug compared to ointment base (vehicle) in subjects with Atopic Dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Diagnosis of atopic dermatitis according to Hanifin and Rajka Criteria
* Willingness of subject to follow all study procedures
* Willingness to avoid excessive exposure of diseased areas to natural or artificial sunlight

Exclusion Criteria:

* Pregnancy and breast-feeding
* Clinically relevant disease, which could interfere with the study conduct or the evaluation and interpretation of the study results
* Clinically manifested immunosuppressive disorder or known history of malignant disease
* History of relevant drug and/or food allergies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Eczema Area and Severity Index (EASI) | Over all study visits for up to 4 weeks

SECONDARY OUTCOMES:
Subjects´ assessment of pruritus | At baseline and after 4 weeks of treatment
  Subjects´ assessment of pruritus using a visual analog scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Berlin, Germany